CLINICAL TRIAL: NCT00929799
Title: Effects of Treatment With Human Growth Hormone on Insulin Resistance and Insulin Secretion in Adults With Growth Hormone Deficiency
Brief Title: Growth Hormone and Glucose Metabolism
Acronym: GHGMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Dr. med AYMAN M. ARAFAT, Charité-University Medicine Berlin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NRA 6280012; EK218-01
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Growth Hormone (Experimental): Therapy with recombinant human GH (Genotropin® 1 mg = 3 IU, Pfizer Inc., NY, USA) daily by subcutaneous injection using a Genotropin pen at maximal GH dose of 0.003 mg/kg/day in patients with severe GHD
  Interventions: Drug: recombinant human Growth Hormone (Genotropin® )

INTERVENTIONS:
Drug: recombinant human Growth Hormone (Genotropin® ) — Once daily by subcutaneous injection using a Genotropin pen in the abdomen at 22:00 h. Maximal GH dose of 0.003 mg/kg/day.

SUMMARY:
The aim of the study is to investigate changes in insulin sensitivity and ß-cell function after 24 and 48 weeks of low-dose growth hormone (GH) therapy in adult patients with severe GH deficiency using highly standardized techniques. Insulin sensitivity was estimated using euglycemic, hyperinsulinemic clamps, while insulin secretion and hepatic insulin clearance were determined by changes in insulin and C-peptide levels during hyperglycemic hyperinsulinemic clamps with consecutive intravenous (i.v.) L-arginine stimulation tests. Moreover, the researchers investigated changes in body composition, lipolysis and cardiovascular risk markers. Furthermore, in order to verify the mechanisms involved in the pathogenesis of GH-induced insulin resistance and the GH-induced improvement in insulin resistance under long term treatment, the researchers intend to establish changes in intramyocellular lipid (IMCL) in patients with GH deficiency by magnetic resonance (MR)-spectroscopy before and during GH-treatment and to correlate IMCL with insulin resistance, insulin secretion and insulin clearance. Finally, the researchers aim to justify the effect of GH on adiponectin secretion as well as on the 11-ß hydroxylase activity.

DETAILED DESCRIPTION:
In adult patients with GH deficiency, it is well documented that treatment with recombinant human GH results in a reduction of visceral fat mass and an increase in muscle mass. During long-term treatment, these effects seem to have beneficial effects on glucose metabolism. However, during the initial phase of GH treatment the insulin antagonistic effect of GH often induces an insulin resistant state which leads to an increase in insulin secretion or even, in cases with a preexisting ß-cell defect, to overt diabetes. Due to the lipolytic effect of GH, an impact of GH treatment on intracellular lipid homeostasis in adipose tissue, but also in skeletal muscle cells and liver cells can be expected. Moreover, since insulin resistance is known to be closely correlated with intramyocellular lipid (IMCL) content, changes in IMCL can play a key role in the GH-induced changes in the insulin sensitivity. Anyway, the mechanisms involved in the pathogenesis of GH-induced insulin resistance and the GH-induced improvement in insulin resistance under long term treatment are presently not fully understood. In order to verify these mechanisms, we intend to establish changes in IMCL in patients with GH deficiency by MR-spectroscopy before and during GH-treatment and to correlate IMCL with insulin resistance, insulin secretion and insulin clearance. Finally, we aim to justify the effect of GH on adiponectin secretion as well as on the 11-ß hydroxylase activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old.
* Severe GH deficiency as diagnosed by an inadequate GH stimulation in three different tests:

  1. peak response < 3 µg/l during an insulin tolerance test;
  2. < 3 µg/l during glucagon test;
  3. < 9 µg/l during GHRH-arginine stimulation test).

Exclusion Criteria:

* GH replacement therapy prior to inclusion.
* History of diabetes Type 1 or 2.
* Biochemical evidence of impaired hepatic or renal function.
* History of cardiovascular disease.
* Uncontrolled hypertension.
* Current inflammatory or malignant disease.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2003-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in insulin sensitivity after 24 and 48 weeks of treatment with low GH dose in severely GH deficient patients. | At 24 and 48 weeks of treatment

SECONDARY OUTCOMES:
Changes from baseline in insulin secretion and insulin clearance, as well as changes in body composition, lipolysis, cardiovascular risk markers, Adiponectin, IMCL and 11ßHSD activity. | At 24 and 48 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ayman M Arafat, Dr.med., Principal Investigator — Charite Campus Benjamin Franklin
Locations (1):
- Charite Campus Benjamin Franklin, Berlin, Germany

REFERENCES:
- [Derived] Arafat AM, Mohlig M, Weickert MO, Schofl C, Spranger J, Pfeiffer AF. Improved insulin sensitivity, preserved beta cell function and improved whole-body glucose metabolism after low-dose growth hormone replacement therapy in adults with severe growth hormone deficiency: a pilot study. Diabetologia. 2010 Jul;53(7):1304-13. doi: 10.1007/s00125-010-1738-4. Epub 2010 Apr 6. PMID 20372873